CLINICAL TRIAL: NCT01125592
Title: Assessment of the Ability of Ionic Foot Bath (IonCleanse®) to Remove Heavy Metals Through the Feet and Its Potential Impact on Body Burden of Heavy Metals
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Responsible Party: Principal Investigator, Dugald Seely, Director of Research & Clinical epidemiology, The Canadian College of Naturopathic Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IonFootbath
Record Dates: First submitted 2010-05-14; First posted 2010-05-18 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: assess the ability of the IonCleanse machine to remove heavy metals through the feet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Footbath (Experimental): Participants in this arm of the study will receive 4 30 minutes ionic footbath sessions, one each week for 4 weeks.
  Interventions: Device: IonCLeanse Footbath

INTERVENTIONS:
Device: IonCLeanse Footbath — Application of an ionic footbath for 30 minutes per week for 4 weeks
  Other Names: IonCleanse SOLO machine manufactured by A Major Difference

SUMMARY:
Makers of ionic foot baths claim that their machines can eliminate heavy metals from the body. Researchers at the Canadian College of Naturopathic Medicine are evaluating the ability of an ionic foot bath to help eliminate heavy metals from the body by rigorously testing the machine under controlled conditions. The machine will first be tested without feet under normal operating conditions and again after operation under normal conditions with foot immersion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adults

Exclusion Criteria:

* A wearer of a pacemaker or any other battery operated or electrical implant
* Pregnant or nursing women
* On heartbeat regulating medication
* On blood thinners (anticoagulants)
* On any drug known to have chelating properties
* Have had an organ transplant or a metal joint implant
* On a medication the absence of which would mentally or physically incapacitate them, e.g., psychotic episodes, seizures, etc.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in heavy metal content in the water after a 30 minute IonCleanse footbath | 4 sessions, May 26 to June 17 2010
  The footbath water will be assessed after each footbath session for each participant via a drinking water assessment performed by an accredited lab.
  Screening for heavy metals will be done via a 24 urine collection and Urine Toxic Metals assessment four times during the study - baseline, during 2nd and 4th footbath sessions and then at the 3 month mark post baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Canadian College of Naturopathic Medicine, Toronto, Ontario, Canada

REFERENCES:
- [Result] Kennedy DA, Cooley K, Einarson TR, Seely D. Objective assessment of an ionic footbath (IonCleanse): testing its ability to remove potentially toxic elements from the body. J Environ Public Health. 2012;2012:258968. doi: 10.1155/2012/258968. Epub 2011 Nov 29. PMID 22174728